CLINICAL TRIAL: NCT03350958
Title: The Impact of Dietary Fibres on Pancreatic Lipase Activity and Gastrointestinal Function
Brief Title: Bioactive Dietary Fibres and Obesity
Acronym: FIBREFOODS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: version 2 14th Feb 2011
Record Dates: First submitted 2017-11-01; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Placebo, controlled double-blind crossover study will recruit participants (males and females, who have previously had ileostomy surgery, but currently have no health issues) from the Newcastle upon Tyne/Gateshead area. Subjects will be randomly allocated to one of two treatment groups. One group will receive a test meal containing the dietary fibre first, then on the second visit, the same meal without dietary fibre. The second group will receive the meal without dietary fibre first, followed by the meal containing dietary fibre on the second visit. For each group, the two visits will be at least 2 weeks apart. As the foods will look exactly the same (the fibres used are colourless and tasteless). As it necessary in double-blind crossover studies, neither the researchers nor the participants will know which food they are receiving at each visit. All randomisation will be carried out in anonymised fashion by an independent researcher, who will code foods and participants accordingly.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As it necessary in double-blind crossover studies, neither the researchers nor the participants will know which food they are receiving at each visit. All randomisation will be carried out in anonymised fashion by an independent researcher, who will code foods and participants accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants received experimental test meal first and placebo comparator meal at the next study visit. Participants to fill out visit questionnaire prior to meal and every 30 minutes thereafter for 5 hours. Samples of ileostomy fluid taken at these time-points, along with blood samples in a subset of participants
  Interventions: Dietary Supplement: Alginate Bread; Other: Control Bread
- Group 2 (Placebo Comparator): Participants received placebo comparator meal first and experimental test meal at the next study visit. Participants to fill out visit questionnaire prior to meal and every 30 minutes thereafter for 5 hours. Samples of ileostomy fluid taken at these time-points, along with blood samples in a subset of participants
  Interventions: Dietary Supplement: Alginate Bread; Other: Control Bread

INTERVENTIONS:
Dietary Supplement: Alginate Bread — 100g Alginate Bread, toasted with 20g of butter.
Other: Control Bread — 100g standard White Bread (control), toasted with 20g of butter.
  Other Names: Standard White bread

SUMMARY:
Obesity is a wide reaching problem in the United Kingdom (UK). The most widely used obesity therapies are based around drugs that reduce dietary fat digestion, and thereby reduce uptake of calories from the diet. While such therapies have proved effective, patient compliance is low due to the unwanted gastrointestinal side effects of these drugs. Dietary fibre is generally classified as dietary material of plant origin that is indigestible to humans. Dietary fibre is in fact a wide range of different compounds that have varied effects on the human body. Initial findings from our laboratory suggest that types of fibre from seaweeds (alginates) can greatly reduce the rate that fat is digested in the laboratory. Our studies have identified which types of fibre are the most effective and our aim is to test whether this reduction in fat digestion is the same within the human body. This will be carried out by sampling the digestive fluid from 40 ileostomy patients over a five hour period following a test meal with and without dietary fibres. All study participants will be provided with test foods specially prepared containing the dietary fibres (e.g. in bread). We will collect data from the participants on what they have eaten and how hungry they feel.

DETAILED DESCRIPTION:
Obesity is a rapidly growing health concern in the Western world. Modifications to diet and lifestyle have been shown to benefit weight loss and weight management, but are often difficult for people to adhere to over a long period. Pharmacological treatments (such as Orlistat the most commonly used anti-obesity drug in the UK) also benefit weight loss, but are expensive to the National Health Service (NHS), and patients often stop taking them due to unwanted gastrointestinal side effect such as diarrhoea and incontinence. Orlistat acts by reducing absorption of dietary fat. Dietary fibre is a term used to describe a divergent range of indigestible compounds of plant origin consumed in the diet that have varied effects on the human body. Recent studies have shown that some types of seaweed dietary fibre (alginates) may act to reduce the rate of fat digestion under similar conditions to the human gut. These fibres have also been easily incorporated into loaves of bread by a local bakers, and were also noted to produce a better tasting product with an increased shelf life. People who tasted the bread were unable to tell it apart from a normal white loaf. Alongside the other better characterised benefits of dietary fibre consumption, such as reduced disease risk and better regularity, these dietary fibres may be an ideal candidate to include in a range of commonly eaten foods as a potential means of reducing dietary fat uptake, and thereby benefitting weight loss and weight maintenance. Within the investigators laboratory studies, assessments of which dietary fibre types are best at reducing fat absorption have been made. The aim is to test the proof of principal that this occurs in the human gut, and that foods incorporating these fibres are well-liked and do not cause unwanted gastrointestinal side effects in two separate participant based studies. This study will test whether the best candidate fibres from the investigators laboratory studies show the ability to reduce fat absorption rates in humans. To do this, the fluid leaving the small intestine of ileostomy patients will be analysed over a five hour period following ingestion of a test meal either with or without the best candidate fibres. Both the researchers and the participants will be blinded as to whether the particular meal the participant is consuming is the one with added fibre or not. The participants will then return at least seven days after the first test meal to consume the other test meal.

Up to 40 free-living adults will be recruited who have previously been through ileostomy surgery at least two years prior to recruitment. Participants will come to the Clinical Research Facility (CRF) and the Royal Victoria Infirmary (RVI) Newcastle for an induction visit, and two separate study visits, at least two weeks apart.

At the induction visit, participants will have a chance to ask the research team members any questions they may have on the study. The research staff member will describe what the participant will have to do within the study in full. A pack will be provided to the participant containing two standard meals and water, which the participant will be asked to consume the night before attending for their two study visits. Informed consent will also be taken at this visit.

Both study visits will be at the same time of day, and will be morning visits (starting 10am or before). The evening before each study visit, participants will consume the standard meal at a set time. The participant will then not have anything else to eat or drink until the study visit (we will provide participants with a bottle of water to drink on the morning of the visit, so that they stay hydrated). At each visit, participants will be provided with a set meal that includes additional dietary fat included (e.g. slices of toast with margarine). At one visit, participants will consume a standard meal, at the other they will consume the same meal with added dietary fibres. Neither the participant nor the researchers will know which meal they are receiving at each visit. These will be randomly labelled and allocated by an independent researcher (who will not have access to participant identifiable information). This type of study is referred to as a double-blind, placebo- controlled trial.

Participants will be asked to fill out questionnaires on their general well-being, abdominal pain and gut health, and feeling of fullness before and after the study meal (every 30 minutes) over a five hour period. At these 30 minute time- points, ileostomy effluent bags will be provided to the participant to replace. The collected effluent will be separated into small vials and anonymised by the researchers. This will then be frozen until it can be analysed later. These samples will be analysed for fat content, carbohydrate content and amount and activity of digestive enzymes and associated compounds (such as bile acids).

At consent, participants will be asked if they would be willing to provide blood samples during the study visits. If they are happy to do this, samples will be taken at hourly intervals over this five hour time period in order to assess the rate of appearance of fats and glucose into the bloodstream. Such samples will be analysed at an accredited Biochemistry laboratory within the hospital. Any results that fall outside of the normal ranges in initial fasting samples will be reported to participants and their General Practitioner (GP) immediately, and participants will be withdrawn from the study. The result of these fasting blood samples will also be sent to both GP and participants following their completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Free-living
* Male or female
* Aged 18 years or above
* Have previously gone through ileostomy surgery at least two years prior, and where the ileostomy procedure is classified as fully functional and stable
* Generally healthy
* Able to fulfill study time commitments and research burden within their usual lifestyle
* In the case of the subset of participants who will give blood samples, that they are happy to provide blood samples

Exclusion Criteria:

* If the original reason for ileostomy (e.g. Crohn's disease, ulcerative colitis or cancer) is active during the study
* Diagnosis of major health issues, either acute or longterm
* Allergy, intolerance of dislike of any study foods

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-03-10 (Actual); Primary Completion 2013-03-07 (Actual); Study Completion 2013-03-07 (Actual)

PRIMARY OUTCOMES:
Measurement of fat excretion in ileostomy effluent | Every 30 minutes for up to 300 minutes after test meal consumption
  Measurement in grams of total lipid in ileal effluent every 30 minutes after test meal consumption

SECONDARY OUTCOMES:
Assessment of general and gut wellbeing | Every 30 minutes for up to 300 minutes after test meal consumption
  Using VAS score from the well being questionnaire
Measurement of circulating triacylglycerol in blood | Every 30 minutes for up to 300 minutes after test meal consumption
  Measured in micro-molar of triacylglycerol (TAG) every 30 minutes after test meal consumption

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.